CLINICAL TRIAL: NCT04076228
Title: Immunophenotyping, Molecular Analysis and Functional Characterization of Cluster of Differentiation Expressing Cells and/or Other Immune Populations in Response to Pembrolizumab in Chinese NSCLC Patients
Brief Title: Biomarkers to Predict the Response to Pembrolizumab in Chinese NSCLC Patients
Status: Completed | Type: Observational
Sponsor: Kiang Wu Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KWH201702
Record Dates: First submitted 2019-08-27; First posted 2019-09-03 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: NSCLC Stage IV
Keywords: NSCLC; PD-L1; Biomarkers
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 7 ml of whole blood from patients and donor will be collected. Blood samples will be stored in EDTA-coating tube. PBMC will be isolated using a density gradient technique. Whole blood will be processed using standard protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pembrolizumab: Chinese lung cancer patients who will receive pembrolizumab will be enrolled in this study. Clinically, the treatment course of pembrolizumab is depended on the efficacy, but average cycle is about 3-4 weeks and patient will receive 6 treatment courses.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — pembrolizumab is a PD-1 inhibitor. Treatment and follow up will be performed at Kiang Wu Hospital in their clinical oncology center. Clinically pathological related information will be recorded.

SUMMARY:
Pembrolizumab is approved for advanced stage non-small cell lung cancer. However, the response rate is low (around 10-15 %) in patients treated in Macau SAR, China. The investigators hypothesize CD38 expressing cells and/or other immune populations will help to predict response.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death, the overall survival rate is low. Recently, using anti-PD-L1 immunotherapy for treatment of cancer shows promising in some types of cancer, including melanoma, head and neck squamous cell cancer, and lung cancer etc. Pembrolizumab is a FDA-approved anti-PD-L1 drug for treatment of advanced stage non-small cell lung cancer. In China, it is approved for used in Macau and Hong Kong. Biomarkers associated with predictive response includes PD-L1 high expression, high mutational burden, and T-cell infiltration based on several clinical trial studies in the western countries. However, the response rate is low (around 10-15 %) in patients treated in Macau SAR, China. The investigators hypothesize that immunophenotying, molecular analysis and functional characterization of CD38 expressing cells and/or other immune populations CD38 will help to identify predictive, Progression and resistance markers associated with PDL1 treatment response. The investigators will collect the blood samples of Pembrolizumab response and non-response Chinese lung cancer patients and compare the imumnophenotypic and molecular dynamic changes during treatment courses. The investigators will also examine the role of CD38 and other molecular markers associated with Pembrolizumab response, functional characterize in vitro. The molecular mechanism controlling Pembrolizumab response will be better understood for designing a better treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Locally advanced (stage IIIB) or metastatic (stage IV) NSCLC, not amenable to curative surgery or radiotherapy
* With PD-L1test available
* Progressed on previous treatment, or treatment native patients. Patients may have also received additional lines of treatment
* Received pembrolizumab treatment in the participating site.

Exclusion Criteria:

* Enrollment in studies that prohibit any participation in this observational study
* No serum samples available

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study cohort will include locally advanced or metastatic NSCLC patients with PD-L1 status available and receive pembrolizumab treatment per the judgement of treating physicians in the participating site in Macau. 30-40 patients are anticipated to be enrolled in the study, the majority of which are estimated to be from mainland China.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Disease response is assessed every 3 weeks for the first 18 weeks and then every 12 weeks until disease progression (worsens) or study completion, an average of 24 months.
  To assess the real world effectiveness of pembrolizumab treatment in locally advanced or metastatic NSCLC patients with PD-L1 positive in terms of response rate

CONTACTS AND LOCATIONS:
Overall Officials: Yabing Cao, MD; PhD, Principal Investigator — Kiang Wu Hospital
Locations (1):
- Kiang Wu Hospital, Macao, China

IPD SHARING:
Plan to Share IPD: No